CLINICAL TRIAL: NCT05972603
Title: Can Topical Vancomycin Prevent Periprosthetic Joint Infection in Primary Hip and Knee Arthroplasty? Multicenter Randomized Controlled Trial
Brief Title: Role of Topical Vancomycin in Reducing Infections in Hip and Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Independent Public Healthcare Center in Rypin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Rheumatoid Arthritis; Avascular Necrosis of Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0,35% povidone-iodine solution lavage (Experimental): 0,35% povidone-iodine solution lavage left in wound for 3 minutes following final implantation.
  Interventions: Procedure: 0,35% povidone-iodine solution lavage
- 1.0 g Vancomycin powder into the wound (Experimental): additional 1.0 g Vancomycin powder into the wound
  Interventions: Procedure: 1.0 g Vancomycin powder into the wound

INTERVENTIONS:
Procedure: 1.0 g Vancomycin powder into the wound — 0,35% povidone-iodine solution lavage left for 3 minutes following final implantation and additional application 1.0 g Vancomycin powder into the wound
  Arms: 1.0 g Vancomycin powder into the wound
Procedure: 0,35% povidone-iodine solution lavage — 0,35% povidone-iodine solution lavage left for 3 minutes following final implantation
  Arms: 0,35% povidone-iodine solution lavage

SUMMARY:
The study is designed to assess the efficacy of vancomycin powder and dilute povidone-iodine lavage (VIP protocol) in reducing the PJI after primary Total Hip Arthroplasty (THA) and Total Knee Arthroplasty (TKA). We hypothesized that VIP protocol provides superior reduction of periprosthetic joint infection (PJI) rates after primary THA and TKA compared with diluted povidone-iodine (PI) protocol.

DETAILED DESCRIPTION:
Patients who undergo primary hip or knee arthroplasty, before closure 0,35% povidone-iodine (17,5mL in 500 mL saline) solution lavage left for 3 minutes following final implantation.

Patients drawn by random numbers calculator will be administered with 1.0 g Vancomycin powder into the wound around the prosthesis and no suction will be used.

ELIGIBILITY:
Inclusion Criteria:

* undergoing THA or TKA as a result of osteoarthritis or rheumatoid arthritis, can understand and comply with the study protocol, have signed the informed consent document at screening

Exclusion Criteria:

* Patients referred to the hospital in order to undergo THA or TKA due to different reason than osteoarthritis, rheumatoid arthritis or avascular necrosis of the femoral head, such as: failed femoral neck fractures, displaced acetabular fractures or revision acetabular fractures, revision knee or hip arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
periprosthetic joint infection | 90 days
  infection rate in each group

CONTACTS AND LOCATIONS:
Locations (1):
- IPHC Rypin, Rypin, Kujawsko-pomorksie, Poland

REFERENCES:
- [Derived] Kulakowski M, Elster K, Szymczak M, Sleczka P, Baumgart M, Krolikowska A, Reichert P. Comparison of the effect of combined usage of povidone-iodine irrigation and topical vancomycin powder to the use of povidone-iodine irrigation alone on the periprosthetic joint infection incidence rate in patients undergoing primary total hip and knee arthroplasty: a protocol for multicenter prospective randomized clinical trial. Trials. 2024 Jul 10;25(1):468. doi: 10.1186/s13063-024-08306-3. PMID 38987786